CLINICAL TRIAL: NCT03840772
Title: ERibulin in Advanced Solitary Fibrous Tumor, an ItaliaN Sarcoma Group Phase II Study (ERASING)
Brief Title: Eribulin in Advanced Solitary Fibrous Tumor
Acronym: ERASING
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISG-ERASING
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Solitary Fibrous Tumor
Keywords: Solitary Fibrous Tumor; soft tissue sarcoma; rare sarcoma
MeSH Terms: conditions — Solitary Fibrous Tumors; Sarcoma | interventions — eribulin

STUDY DESIGN:
Intervention Model Description: Not controlled, single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eribulin (Experimental): Eribulin will be administered at the dose of 1.23 mg/m², intravenously over 2-5 min on day 1 and day 8 of every 21 day cycle.
  Study treatment will be administered until evidence of progression or unacceptable toxicity, patient's own willingness, non-compliance or according to clinical investigator's decision.
  Interventions: Drug: Eribulin

INTERVENTIONS:
Drug: Eribulin — Treatment with eribulin
  Other Names: Intervention under investigation

SUMMARY:
Phase II study on advanced Solitary Fibrous Tumor (SFT) treated with eribulin

DETAILED DESCRIPTION:
This is an Italian, non randomized, open label, multi center, investigator-initiated, Phase II, clinical study to explore the activity of eribulin in a population of patients with progressive, advanced (i.e. locally advanced or metastatic), molecularly proven SFT. Patients with a documented and centrally reviewed pathological diagnosis of locally advanced or metastatic SFT, and with an evidence of progression within the previous 6 months, may enter the study.

Study treatments will be administered till progression or toxicity. The primary end-point of the study is overall response rate Secondary end-points are Progression Free Survival (PFS), Overall Survival (OS) clinical benefit rate, response rate as by Choi criteria, duration of response.

Subjects already treated with one or two prior medical therapy regimens for the advanced phase, whatever agent used in first- or second-line, are eligible for inclusion in the study. Investigators will consider eligible for this study even patients naïve from chemotherapy, considering the limited activity of anthracycline in the disease.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or legal representative must be able to read and understand the informed consent form and must have been willing to give written informed consent and any locally required authorization before any study-specific procedures, including screening evaluations, sampling, and analyses
2. Age ≥18 years
3. Histological centrally and molecular confirmed diagnosis SFT
4. Locally advanced disease and/or metastatic disease
5. Measurable disease according RECIST 1.1
6. Evidence of progression by RECIST 1.1 during the 6 months before study entry
7. Patients must be treated with at least one prior medical anticancer treatment line for the advanced phase of disease (both cytotoxic chemotherapy or target treatment allowed) and with a maximum of 2 lines.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
9. Adequate bone marrow function
10. Adequate organ function
11. Cardiac ejection fraction ≥50%
12. Female patients of child-bearing potential must have negative pregnancy test within 7 days before initiation each cycle of chemotherapy. Post-menopausal women must be amenorrhoeic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective method of birth control throughout the study.

Exclusion Criteria:

1. Naïve patients
2. More than 2 lines of anticancer treatment
3. Previous treatment with any other anti-cancer investigational or not investigational agents within 21 days of first day of study drug dosing,
4. Previous treatment with radiation therapy within 14 days of first day of study drug dosing, or patients who have not recovered from adverse events due to agents previously administered
5. Previous radiotherapy to 25% of the bone marrow
6. Major surgery within 21 days prior to study entry
7. Other primary malignancy with <5 years clinically assessed disease-free interval, except basal cell skin cancer, cervical carcinoma in situ, or other neoplasms judged to entail a low risk of relapse
8. Pregnancy or breast feeding
9. Cardiovascular diseases resulting in a New York Heart Association Functional Status >2 . Medical history of a myocardial infarction < 6 months prior to initiation of study treatment. Unstable angina or myocardial infarction within 6 months of enrolment, Serious and potentially life-threatening arrhythmia
10. Subjects with a high probability of Long QT Syndrome or corrected QT interval prolongation of more than or equal to 501 msec , following correction of any electrolyte imbalance
11. Medical history of arterial thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), or pulmonary embolism within 6 months prior to the initiation of study treatment
12. Known history of human immunodeficiency virus infection
13. Active or chronic hepatitis B or C requiring treatment with antiviral therapy
14. Medical history of hemorrhage or a bleeding event ≥ Grade 3 according Common Terminology Criteria for Adverse Events (CTCAE) within 4 weeks prior to the initiation of study treatment
15. Evidence of any other serious or unstable illness, or medical, psychological, or social condition, that could jeopardize the safety of the subject and/or his/her compliance with study procedures, or may interfere with the subject's participation in the study or evaluation of the study results
16. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation of the study drugs
17. Subjects who have not recovered from acute toxicities as a result of prior anti-cancer therapy to ≤ Grade 1 of CTCAE, except for peripheral neuropathy and alopecia.
18. Pre-existing peripheral neuropathy > CTCAE Grade 2.
19. Expected non-compliance to medical regimens
20. Subjects with known central nervous system metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
RECIST 1.1 Overall response rate | At week 6
  Proportion of patients with tumor size reduction ⩾ to 30% measured with RECIST Criteria 1.1

SECONDARY OUTCOMES:
Choi Response Rate | At week 6
  Proportion of patients with tumor size reduction ⩾10% or a decrease in tumour attenuation⩾15% measured with Choi criteria
Overall Survival (OS) at 3 years | At 3 years
  Survival from the first eribulin dose to death for any cause
Progression Free Survival (PFS) at 3 years | At 3 years
  Survival without disease progression
Clinical Benefit Rate | At week 18
  Proportion of patients with no disease progression after 18 weeks of therapy.
Safety of the treatment in term of adverse event | Week 9, week 18, week 27, week 36
  Safety in term of adverse event is evaluate from the first eribulin dose throughout the study according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Stacchiotti, MD, Principal Investigator — Fondazione IRCCS INT di Milano
Locations (3):
- Italy (3):
  - Azienda Ospedaliera Universitaria Paolo Giaccone, Palermo, PA
  - Policlinico Universitario Campus Biomedico, Roma, RM
  - Fondazione IRCCS INT Milano, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verbeke SL, Fletcher CD, Alberghini M, Daugaard S, Flanagan AM, Parratt T, Kroon HM, Hogendoorn PC, Bovee JV. A reappraisal of hemangiopericytoma of bone; analysis of cases reclassified as synovial sarcoma and solitary fibrous tumor of bone. Am J Surg Pathol. 2010 Jun;34(6):777-83. doi: 10.1097/PAS.0b013e3181dbedf1. PMID 20421780
- [Background] Robinson DR, Wu YM, Kalyana-Sundaram S, Cao X, Lonigro RJ, Sung YS, Chen CL, Zhang L, Wang R, Su F, Iyer MK, Roychowdhury S, Siddiqui J, Pienta KJ, Kunju LP, Talpaz M, Mosquera JM, Singer S, Schuetze SM, Antonescu CR, Chinnaiyan AM. Identification of recurrent NAB2-STAT6 gene fusions in solitary fibrous tumor by integrative sequencing. Nat Genet. 2013 Feb;45(2):180-5. doi: 10.1038/ng.2509. Epub 2013 Jan 13. PMID 23313952
- [Background] Dagrada GP, Spagnuolo RD, Mauro V, Tamborini E, Cesana L, Gronchi A, Stacchiotti S, Pierotti MA, Negri T, Pilotti S. Solitary fibrous tumors: loss of chimeric protein expression and genomic instability mark dedifferentiation. Mod Pathol. 2015 Aug;28(8):1074-83. doi: 10.1038/modpathol.2015.70. Epub 2015 May 29. PMID 26022454
- [Background] Chamberlain MC, Glantz MJ. Sequential salvage chemotherapy for recurrent intracranial hemangiopericytoma. Neurosurgery. 2008 Oct;63(4):720-6; author reply 726-7. doi: 10.1227/01.NEU.0000325494.69836.51. PMID 18981882
- [Background] Galanis E, Buckner JC, Scheithauer BW, Kimmel DW, Schomberg PJ, Piepgras DG. Management of recurrent meningeal hemangiopericytoma. Cancer. 1998 May 15;82(10):1915-20. PMID 9587125
- [Background] Beadle GF, Hillcoat BL. Treatment of advanced malignant hemangiopericytoma with combination adriamycin and DTIC: a report of four cases. J Surg Oncol. 1983 Mar;22(3):167-70. doi: 10.1002/jso.2930220306. PMID 6682161
- [Background] Stacchiotti S, Libertini M, Negri T, Palassini E, Gronchi A, Fatigoni S, Poletti P, Vincenzi B, Dei Tos AP, Mariani L, Pilotti S, Casali PG. Response to chemotherapy of solitary fibrous tumour: a retrospective study. Eur J Cancer. 2013 Jul;49(10):2376-83. doi: 10.1016/j.ejca.2013.03.017. Epub 2013 Apr 6. PMID 23566418
- [Background] Schoffski P, Chawla S, Maki RG, Italiano A, Gelderblom H, Choy E, Grignani G, Camargo V, Bauer S, Rha SY, Blay JY, Hohenberger P, D'Adamo D, Guo M, Chmielowski B, Le Cesne A, Demetri GD, Patel SR. Eribulin versus dacarbazine in previously treated patients with advanced liposarcoma or leiomyosarcoma: a randomised, open-label, multicentre, phase 3 trial. Lancet. 2016 Apr 16;387(10028):1629-37. doi: 10.1016/S0140-6736(15)01283-0. Epub 2016 Feb 10. PMID 26874885
- [Background] Schoffski P, Ray-Coquard IL, Cioffi A, Bui NB, Bauer S, Hartmann JT, Krarup-Hansen A, Grunwald V, Sciot R, Dumez H, Blay JY, Le Cesne A, Wanders J, Hayward C, Marreaud S, Ouali M, Hohenberger P; European Organisation for Research and Treatment of Cancer (EORTC) Soft Tissue and Bone Sarcoma Group (STBSG). Activity of eribulin mesylate in patients with soft-tissue sarcoma: a phase 2 study in four independent histological subtypes. Lancet Oncol. 2011 Oct;12(11):1045-52. doi: 10.1016/S1470-2045(11)70230-3. Epub 2011 Sep 19. PMID 21937277
- [Background] Kawai A, Araki N, Naito Y, Ozaki T, Sugiura H, Yazawa Y, Morioka H, Matsumine A, Saito K, Asami S, Isu K. Phase 2 study of eribulin in patients with previously treated advanced or metastatic soft tissue sarcoma. Jpn J Clin Oncol. 2017 Feb 1;47(2):137-144. doi: 10.1093/jjco/hyw175. PMID 28173193
- [Background] Van Glabbeke M, Verweij J, Judson I, Nielsen OS; EORTC Soft Tissue and Bone Sarcoma Group. Progression-free rate as the principal end-point for phase II trials in soft-tissue sarcomas. Eur J Cancer. 2002 Mar;38(4):543-9. doi: 10.1016/s0959-8049(01)00398-7. PMID 11872347